CLINICAL TRIAL: NCT03964207
Title: A Randomized, Open-label, Two-way Crossover Study to Compare Patient Acceptability/Preference of Tiotropium Respimat® With Tiotropium Handihaler® in Patients With Moderate to Very Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study on Whether Patients Prefer the Spiriva® Respimat® or the Spiriva® Handihaler® for Treating Their Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0205-0541
Record Dates: First submitted 2019-05-24; First posted 2019-05-28 (Actual); Results first posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (T1): 5μg tiotropium Respimat®, then (T2): 18μg tiotropium Handihaler® (Experimental): From Day 1 of Period 1 participants received Test treatment (T1): tiotropium Respimat® (Spiriva® Respimat®) 5 microgram (μg) once daily for a duration of 4 weeks, given as 2.5μg per puff, two puffs (2.5μg per puff) inhalation solution of tiotropium, orally via Respimat®.
  From Day 1 of Period 2 participants received comparator treatment(T2): tiotropium Handihaler® (Spiriva®) 18μg once daily for a duration of 4 weeks, inhalation powder tiotropium with 1 Handihaler® device.
  Interventions: Drug: Tiotropium Respimat® (T1); Drug: Tiotropium Handihaler® (T2)
- (T2): 18μg tiotropium Handihaler®, then (T1): 5μg tiotropium Respimat® (Experimental): From Day 1 of Period 1 participants received comparator treatment (T2): tiotropium Handihaler® (Spiriva®) 18 microgram (μg) once daily for a duration of 4 weeks, inhalation powder tiotropium with 1 Handihaler® device.
  From Day 1 of Period 2 participants received Test treatment (T1): tiotropium Respimat® (Spiriva® Respimat®) 5 microgram (μg) once daily for a duration of 4 weeks, given as 2.5μg per puff, two puffs (2.5μg per puff) inhalation solution of tiotropium, orally via Respimat®.
  Interventions: Drug: Tiotropium Respimat® (T1); Drug: Tiotropium Handihaler® (T2)

INTERVENTIONS:
Drug: Tiotropium Respimat® (T1) — inhalation solution
Drug: Tiotropium Handihaler® (T2) — Inhalation Powder

SUMMARY:
The objective of this study is to investigate the patient acceptability/preference of Respimat® compared with Handihaler® in patients with moderate to very severe chronic obstructive pulmonary disease (COPD) to demonstrate the superiority of Respimat®.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of COPD and must meet the following spirometric criteria at Visit 1 (Screening).

  * Relatively stable, moderate to very severe airway obstruction with a post-bronchodilator FEV1 <80% of predicted normal and FEV1/FVC <70%. Spirometry should be done at baseline and approximately 1/2 hour following 4 inhalations of albuterol.
  * Male = exp [-10.61669 + 2.27078 × ln (- in cm) + 0.06622 × ln (age in year) + Mspline] Female = exp [-9.69716 + 2.09385 × ln (- in cm) + 0.02006 × ln (age in year) + Mspline]
  * Historical data from spirometry measurements within the past 6 either at the site or at the other hospital may be used. If the measurements are not performed at the trial site a referral letter and signed copies of the measurement printouts must be provided to the trial site for source data verification. In case several qualifying spirometry measurements are available, the most recent one should be referred to as long as it was not performed during an exacerbation. Patients may not be randomised to the study without the availability of spirometry data at the actual study site.
* Male or female, age: ≥40 years of age
* Patients must be current or ex-smokers with a smoking history of ≥ 10 pack years. (Patients who have never smoked cigarettes must be excluded).
* Signed and dated written informed consent in accordance with International Council on Harmonization (ICH) ICH-GCP and local legislation prior to admission to the trial
* Patients must be able to inhale medication from the Tiotropium Respimat® and Tiotropium HandiHaler®
* Patients must be able to perform all study related procedures, and must be able to maintain records (patient diary) during the study period as required by the protocol

Exclusion Criteria:

* Had visual, cognitive, or motor impairment that, as judged by the investigator, did not allow the patient to independently read and complete the PASAPQ questionnaire
* Patients have had used both Respimat® and HandiHaler® (including generic HandiHaler®) within one year prior to screening.
* Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease or condition which, in the opinion of the investigator, may put the patients at risk because of participation in the study or may influence either the results of the study or the patient's ability to participate in the study.
* All patients with an Aspartate Transaminase (AST) (serum glutamic-oxaloacetic transaminase, SGOT) >80 IU/L, Alanine Aminotransferase (ALT) (Serum Glutamic-pyruvic Transaminase, SGPT) >80 IU/L, Bilirubin >2.0 mg/dL or Creatinine >2.0 mg/dL will be excluded regardless of the clinical condition. Repeat laboratory evaluation will not be conducted in these subjects.
* Patients with a recent history (i.e., one year or less) of myocardial infarction.
* Patients who have been hospitalized or being treated for heart failure within the past year.
* Patients with any unstable or life-threatening cardiac arrhythmia requiring intervention or change in drug therapy during the last year.
* Patients with a malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years (patients with treated basal cell carcinoma are allowed).
* Known active tuberculosis.
* Patients with a history of asthma, cystic fibrosis, clinically not well-controlled bronchiectasis, interstitial lung disease, or pulmonary thromboembolic disease
* History of thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated.
* Patients with any respiratory tract infection or COPD exacerbation in the 6 weeks prior to the initial screening visit (Visit 1).
* Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction. Patients whose symptoms are controlled on treatment may be included.
* Patients with known narrow-angle glaucoma
* Use of systemic corticosteroid medication at unstable doses (i.e., less than six weeks on stable dose) or at doses in excess of the equivalent of 10 milligrams (mg) prednisolone per day.
* Patients who regularly use daytime oxygen therapy for more than 1 hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy.
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e., oral or injectable contraceptives, intrauterine devices (IUD) or diaphragm with spermicide, or Norplant®).
* Significant alcohol or drug abuse within the past 12 months
* Known hypersensitivity to anticholinergic drugs, lactose, benzalkonium chloride (BAC), ethylenediaminetetraacetic acid (EDTA) or any other components of the HandiHaler® or Respimat® inhalation solution delivery system.
* Patients currently in any pulmonary rehabilitation program or scheduled to participate in any such program during the study period.
* Previous participation in this study. (The patient cannot re-enroll into this study.)
* Patients who are currently participating in another interventional study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-11-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Beijing Chao-Yang Hospital, Beijing
  - China-Japan Friendship Hospital, Beijing
  - West China Hospital, Chengdu
  - The First Afiliated Hospital, Sun Yet-sen University, Guangzhou
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - The First Hospital of China Medical University, Shenyang

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, open-label, 2 -way cross-over design, to compare patient acceptability/preference of Tiotropium Respimat® (T1),with Tiotropium Handihaler® (T2) in patients with moderate to very severe chronic obstructive pulmonary disease (COPD).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: First Treatment
Arm/Group | (T1): 5μg Tiotropium Respimat®, Then (T2): 18μg Tiotropium Handihaler® | (T2): 18μg Tiotropium Handihaler®, Then (T1): 5μg Tiotropium Respimat®
Started (Randomized) | 37 | 35
Treated | 36 | 35
Completed | 34 | 33
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Second Treatment
Arm/Group | (T1): 5μg Tiotropium Respimat®, Then (T2): 18μg Tiotropium Handihaler® | (T2): 18μg Tiotropium Handihaler®, Then (T1): 5μg Tiotropium Respimat®
Started | 34 | 33
Completed | 33 | 30
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Population: Treated set (TS) is defined as all patients who were dispensed study medication and were documented to have at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | (T1): 5μg Tiotropium Respimat®, Then (T2): 18μg Tiotropium Handihaler® | (T2): 18μg Tiotropium Handihaler®, Then (T1): 5μg Tiotropium Respimat® | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.4 (6.54) | 65.2 (7.23) | 66.3 (6.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 34 | 35 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 36 | 35 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 36 | 35 | 71
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Performance Domain of the Patient Satisfaction and Preference Questionnaire (PASAPQ) After 4 Weeks of Treatment
Description: The score on the performance domain of the Patient satisfaction and preference questionnaire (PASAPQ) after 4 weeks of treatment is reported. The performance domain score is the sum of 7 questions (Q) within the domain (Q1, Q2, Q3, Q4, Q5, Q10 and Q11), the range for each question went from 1 to 7 the higher the better. The score was then transformed to a 0 (least) to 100 (most) point scale following ((Q1+Q2+Q3+Q4+Q5+Q10+Q11)/49)*100, the higher the better performance. The performance domain of PASAPQ) was analysed using Mixed-effects Model for Repeated Measures (MMRM), with treatment and period as fixed effects, and patient as a random effect. Compound symmetry was used as a covariance structure for within-patient variation.
Time Frame: After 4 weeks of treatment (at week 4 and week 8)
Population: Full analysis set (FAS) is defined as all patients who were randomized to treatment sequence and received at least one dose of one study drug and providing at least one PASAPQ score measurement. Only patients with no missing values were included for the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- (T1): 5μg Tiotropium Respimat®: Participants received Test treatment (T1): tiotropium Respimat® (Spiriva® Respimat®) 5 microgram (μg) once daily for a duration of 4 weeks, given as 2.5μg per puff, two puffs (2.5μg per puff) inhalation solution of tiotropium, orally via Respimat®.
- (T2): 18μg Tiotropium Handihaler®: Participants received comparator treatment (T2): tiotropium Handihaler® (Spiriva®) 18 microgram (μg) once daily for a duration of 4 weeks, inhalation powder tiotropium with 1 Handihaler® device.
Arm/Group | (T1): 5μg Tiotropium Respimat® | (T2): 18μg Tiotropium Handihaler®
Number analyzed (Participants) | 66 | 68
Scores on a scale | 79.830 (15.052) | 85.112 (11.583)
Statistical Analysis 1: Comparison: (T1): 5μg Tiotropium Respimat® vs (T2): 18μg Tiotropium Handihaler®; The hypothesis test was held to investigate the superiority of the test treatment. Mixed-effects Model for Repeated Measures (MMRM) was used to analyze the performance domain of PASAPQ score, with treatment and period as fixed effects, and patient as a random effect; Test type: Superiority; p = 0.007, Mixed-effects Model; Difference of LSmeans = -5.28, 95% CI 2-sided [-9.07 to -1.48] — The Least squares means (LSmeans) were adjusted with treatment and visit. And the Difference of LSmeans was calculated as: value from the test treatment group - value from the comparator treatment group

2. Secondary Outcome: PASAPQ Total Score After 4 Weeks of Treatment
Description: The total score on the Patient satisfaction and preference questionnaire (PASAPQ) after 4 weeks of treatment is reported. The Total score is the sum of 13 questions (Q1-Q13) and then transformed to a 0 (least) to 100 (most) point scale. This continuous secondary endpoint was analyzed using a similar MMRM model as for the primary endpoint.
Time Frame: After 4 weeks of treatment (at week 4 and week 8)
Population: Full analysis set (FAS) is defined as all patients who were randomized to treatment sequence and received at least one dose of one study drug and providing at least one PASAPQ score measurement. Only participants with non-missing results were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | (T1): 5μg Tiotropium Respimat® | (T2): 18μg Tiotropium Handihaler®
Number analyzed (Participants) | 66 | 68
Scores on a scale | 81.51 (13.67) | 85.69 (10.802)
Statistical Analysis 1: Comparison: (T1): 5μg Tiotropium Respimat® vs (T2): 18μg Tiotropium Handihaler®; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.024, Mixed Models Analysis; Difference of LSmeans = -4.14, 95% CI 2-sided [-7.72 to -0.56] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Patients Indicating Preference at Week 8
Description: The percentage of patients indicating preference in the Patient satisfaction and preference questionnaire (PASAPQ) at week 8 is reported. The questionnaire PASAPQ is a two part questionnaire, in Part II of the PASAPQ the stand-alone question 15 (Q15) was asked for a response to indicate the preference for the trial device, it had three possible answers: "I prefer Respimat", "I prefer Handihaler", "No answer to this question " and "no preference". Chi-squared test was used to analyze proportion of patients indicating preference in the Patient satisfaction and preference questionnaire (PASAPQ) at week 8.
Time Frame: At Week 8.
Population: Full analysis set (FAS) is defined as all patients who were randomized to treatment sequence and received at least one dose of one study drug and providing at least one PASAPQ score measurement.
Measure: Number; unit: Percentage
Groups:
- Tiotropium (T1 or T2): Participants received Test treatment: 5μg tiotropium Respimat® (T1) or 18μg tiotropium Handihaler® (T2):
  Tiotropium Respimat® (Spiriva® Respimat®) 5 microgram (μg) once daily for a duration of 4 weeks, given as 2.5μg per puff, two puffs (2.5μg per puff) inhalation solution of tiotropium, orally via Respimat®.
  Tiotropium Handihaler® (Spiriva®) 18 microgram (μg) once daily for a duration of 4 weeks, inhalation powder tiotropium with 1 Handihaler® device.
Arm/Group | Tiotropium (T1 or T2)
Number analyzed (Participants) | 69
Percentage
  I prefer Respimat | 50.7
  I prefer Handihaler | 37.7
  No preference | 5.8
  No answer to this question | 5.8
Statistical Analysis 1: Comparison: Tiotropium (T1 or T2); Chi-squared test was used to analyze proportion of patients indicating preference in the Patient satisfaction and preference questionnaire (PASAPQ) at week 8. All participants have used both treatments at this point: Handihaler (4 weeks) and Respimat (4 weeks); Test type: Superiority; p = 0.249, Chi-square test; Difference rate (%) = 13.0 — The Difference rate was calculated as: value from the test treatment group - value from the comparator treatment group

4. Secondary Outcome: Overall Satisfaction Question Score From PASAPQ After 4 Weeks of Treatment
Description: The overall satisfaction question score in the Patient satisfaction and preference questionnaire (PASAPQ) at week 4 and 8 is reported (after 4 weeks of treatment). In Part I of the questionnaire PASAPQ: the Question 14 (Q14) asked for the overall satisfaction with the device used in the study. Q14 had Likert-type response options of 1 (very dissatisfied) to 7 (very satisfied) and was then transformed to a 0 (least) to 100 (most) point scale (if a patient scored "x", the transfer to 0-100 scale was x/7*100). Mixed-effects Model for Repeated Measures (MMRM) was used to analyze the overall satisfaction question score, with treatment and period as fixed effects, and patient as a random effect.
Time Frame: At the end of 4 weeks of treatment
Population: Full analysis set (FAS) is defined as all patients who were randomized to treatment sequence and received at least one dose of one study drug and providing at least one PASAPQ score measurement. Only participants with non-missing endpoints were included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | (T1): 5μg Tiotropium Respimat® | (T2): 18μg Tiotropium Handihaler®
Number analyzed (Participants) | 66 | 68
Score on a scale | 82.56 (19.702) | 87.24 (12.257)
Statistical Analysis 1: Comparison: (T1): 5μg Tiotropium Respimat® vs (T2): 18μg Tiotropium Handihaler®; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.057, The mixed model for repeated measures; Difference of LSmeans = -4.72, 95% CI 2-sided [-9.59 to 0.15] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Score on Willingness to Continue at Week 8
Description: The score on willingness to continue in the Patient satisfaction and preference questionnaire (PASAPQ) at week 8 is reported. The PASAPQ is a two part questionnaire, in Part I of the questionnaire PASAPQ the Question 16 (Q16) asked for a response between 0 and 100 with 0 indicating not willing to continue using the trial device and 100 indicating definitely willingness to continue. Mixed-effects Model for Repeated Measures (MMRM) was used to analyze the score on willingness to continue, with treatment and period as fixed effects, and patient as a random effect.
Time Frame: At Week 8.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | (T1): 5μg Tiotropium Respimat® | (T2): 18μg Tiotropium Handihaler®
Number analyzed (Participants) | 65 | 65
Scores on a scale | 82.9 (28.10) | 87.3 (19.19)
Statistical Analysis 1: Comparison: (T1): 5μg Tiotropium Respimat® vs (T2): 18μg Tiotropium Handihaler®; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.347, Mixed Models Analysis; Difference of LSmeans = -4.38, 95% CI 2-sided [-13.63 to 4.86] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first treatment intake until 28 days after last treatment intake. Up to 56 days.
Description: Treated set (TS) is defined as all patients who were dispensed study medication and were documented to have at least one dose of investigational treatment.
Arm/Group | (T1): 5μg Tiotropium Respimat® | (T2): 18μg Tiotropium Handihaler®
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/69
Serious Adverse Events (participants affected / at risk) | 2/69 | 2/69
Other Adverse Events (participants affected / at risk) | 0/69 | 0/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | (T1): 5μg Tiotropium Respimat® (N=69) | (T2): 18μg Tiotropium Handihaler® (N=69)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT03964207/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT03964207/SAP_001.pdf